CLINICAL TRIAL: NCT01059344
Title: A Randomized Placebo-Controlled Double-Blind Study to Evaluate the Efficacy and Safety of Asacol™ 4.8 g/Day (800 mg Tablets) for the Treatment of Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Asacol™ 4.8 g/Day (800 mg Tablets) for the Treatment of Active Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP0203
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Ulcerative Colitis
Keywords: Mesalamine; Asacol; Ulcerative colitis; induction therapy; acute disease; mild to moderate; Active Ulcerative Colitis (mild to moderate)
MeSH Terms: conditions — Colitis, Ulcerative; Acute Disease | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesalamin (Experimental): 4.8g Mesalamin (800mg tablet)
  Interventions: Drug: Mesalamin
- Placebo (Placebo Comparator): 4.8g Placebo to Mesalamin (800 mg tablet)
  Interventions: Drug: Mesalamin

INTERVENTIONS:
Drug: Mesalamin — 4.8g/day, 800 mg tablets
  Other Names: Asacol

SUMMARY:
The primary objective of the study is to determine the efficacy of Asacol™ 4.8 g/day (800 mg tablets) to induce clinical and endoscopic remission after 6 weeks of treatment compared to placebo in subjects with active ulcerative colitis (UC).

DETAILED DESCRIPTION:
The 800 mg Asacol™ tablets from Tillotts Pharma AG are being marketed in over 30 countries, mainly in Europe and Asia. Approved dosages for the treatment of active UC are between 2.4 and 4.8 g/day in analogy to the approved 400 mg dosage form. The present trial is planned to generate efficacy data to support the safe use of a 4.8 g/day dose of the 800 mg dosage form in a well defined population of patients with mildly to moderately active UC. In keeping with the EMEA UC guideline the study will have a placebo-controlled 6 weeks induction treatment. After 6 weeks, treatment success will be evaluated using the modified UC disease activity index as primary efficacy measurement.

ELIGIBILITY:
Inclusion Criteria:

(1) Male or non-pregnant, non-lactating females, 18 years of age or older. (2) Documented diagnosis of UC with disease extending at least 15 cm from the anal verge.

(3) Active UC defined by:

(a) modified UC-DAI score of 4-10 with (b) sigmoidoscopy component score ≥ 2 and (c) rectal bleeding component score ≥ 1 (4) Ability of subject to participate fully in all aspects of this clinical trial.

(5) Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Severe UC defined by the following criteria:

   ³6 bloody stools daily with one or more of the following:
   1. oral temperature > 37.8°C or > 100.0°F
   2. pulse > 90/min
   3. hemoglobin < 10 g/dL
2. Previously failed treatment with a mesalazine dose of > 2.0 g/day.
3. Current relapse lasting > 6 weeks in the opinion of the investigator.
4. Treatment with 5-ASA at a dose of >2.0g/day within 1 week prior to randomisation
5. Treatment with systemic or rectal steroids within 4 weeks prior to randomization.
6. Treatment with immunosuppressants within 6 weeks prior to randomization.
7. Treatment with infliximab or other biologics within 3 months prior to randomization.
8. Treatment with systemic antibiotics for UC within 7 days prior to randomization.
9. Treatment with probiotics within 7 days prior to randomization.
10. Treatment with anti-diarrheals within 7 days prior to randomization.
11. Treatment with nicotine patch within 7 days prior to randomization.
12. Received any investigational drug within 30 days prior to randomization.
13. History of colectomy or partial colectomy.
14. History of definite dysplasia in colonic biopsies.
15. Crohn's disease.
16. Known bleeding disorders.
17. Immediate or significant risk of toxic megacolon.
18. Hypersensitivity to salicylates, aspirin, sulfasalazine or 5-ASA.
19. Serum creatinine > 1.5 times the upper limit of the normal range.
20. AST, ALT, total bilirubin or alkaline phosphatase > 2 times the upper limit of the normal range.
21. Serious underlying disease other than UC which in the opinion of the investigator may interfere with the subject's ability to participate fully in the study.
22. History of alcohol or drug abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.
23. Stools positive for clostridium difficile.
24. Pregnant or lactating women.
25. Prior enrolment in the current study and had received study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Feagan, MD, Study Chair — Alimentiv Inc.
Locations (31):
- Belarus (6):
  - Gomel Regional Clinical Hospital, 9, Homyel
  - City Clinical Hospital No.1, Minsk
  - Minsk Regional Clinical Hospital, 41, Minsk
  - City Clinical Hospital No. 2, Minsk
  - E.Klumov City Clinical Hospital No. 3, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- India (8):
  - Medwin Hospital, Hyderabad, Andhrapradesh
  - Osmania General Hospital, Hyderabad, Andhrapradesh
  - M.S.Ramiah Hospital, Bangalore, Karnataka
  - Shree Gokulam Medical College and Research Foundation, Trivandrum, Kerala
  - S. R. Kalla Memorial Gastro and General Hospital, Jaipur, Rajasthan
  - Life Line Hospital, Chennai, Tamil Nadu
  - Maulana Azad Medical College and Associated Lok Nayak Hospital, New Delhi
  - Institute of liver and billiary sciences, New Delhi
- Turkey (Türkiye) (9):
  - Ankara University Medical Faculty Sihhiye, Ankara
  - Hacettepe University Medical Faculty Sihhiye, Ankara
  - Gazi University Medical Faculty Besevler, Ankara
  - Dicle University Medical Faculty, Diyarbakır
  - Trakya University Medical Faculty, Edirne
  - Gaziantep University Medical Faculty Kampus Alani, Gaziantep
  - Sisli Etfal Egitim ve Arastirma Hospital Sisli, Istanbul
  - Dokuz Eylul University Medical Faculty Inciralti, Izmir
  - Ataturk Egitim ve Arastirma Hospital Basin Sitesi, Izmir
- Ukraine (8):
  - Dnipropetrovska derzhavna medychna akademiia,, Dnipropetrovsk
  - Ivano-Frankivskyi natsionalnyi medychnyi universytet,, Ivano-Frankivsk
  - Miska klinichna likarnia 2,, Kharkiv
  - Natsionalnyi medychnyi universytet im. Bogomoltsia, kafedra khirurgii 1 na bazi viddilennia proctologii Miskoi klinichnoi likarni 18, m.Kyiv, Kyiv
  - Natsionalnyi medychnyi universytet im. O.O. Bogomoltsia,, Kyiv
  - Natsionalna medychna akademia pisliadyplomnoi osvity im. P.L. Shupyk,, Kyiv
  - Lvivskyi natsionalnyi medychnyi universytet imeni Danyla Galytskogo,, Lviv
  - Odeska oblasna klinichna likarnia, Oblasnyi tsentr gastroenterologii,, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feagan BG, Sandborn WJ, D'Haens G, Pola S, McDonald JWD, Rutgeerts P, Munkholm P, Mittmann U, King D, Wong CJ, Zou G, Donner A, Shackelton LM, Gilgen D, Nelson S, Vandervoort MK, Fahmy M, Loftus EV Jr, Panaccione R, Travis SP, Van Assche GA, Vermeire S, Levesque BG. The role of centralized reading of endoscopy in a randomized controlled trial of mesalamine for ulcerative colitis. Gastroenterology. 2013 Jul;145(1):149-157.e2. doi: 10.1053/j.gastro.2013.03.025. Epub 2013 Mar 22. PMID 23528626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2009 - February 2011
Pre-assignment Details: Screen failures, not complying to inclusion and exclusion criteria
Groups:
- Placebo: Placebo to Mesalamin: 4.8g/day, 800 mg tablets
Period: Overall Study
Arm/Group | Mesalamin | Placebo
Started | 140 | 141
Completed | 118 | 95
Not Completed | 22 | 46
Not completed — Adverse Event | 12 | 30
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Lost to Follow-up | 1 | 1
Not completed — Other | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Mesalamin: Mesalamin: 4.8g/day, 800 mg tablets The study drug will be given for 10 weeks. All treatment regimens will be orally administered, with or without food. Subjects randomized to the Asacol™ 4.8 g/day treatment group will receive three 800 mg Asacol™ tablets in the morning and three 800 mg Asacol™ tablets in the evening.
- Placebo: Placebo to Mesalamin: 4.8g/day, 800 mg tablets The study drug will be given for 10 weeks. All treatment regimens will be orally administered, with or without food. Subjects randomized to the placebo treatment group will receive three placebo tablets in the morning and three placebo tablets in the evening.
- Total: Total of all reporting groups
Arm/Group | Mesalamin | Placebo | Total
Number analyzed (Participants) | 140 | 141 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (14.3) | 40.72 (13.8) | 41.8 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 66 | 119
  Male | 87 | 75 | 162
Race/Ethnicity, Customized [Number; unit: participants]
  White | 114 | 110 | 224
  Asian | 26 | 31 | 57
Region of Enrollment [Number; unit: participants]
  Turkey | 13 | 11 | 24
  Ukraine | 54 | 55 | 109
  Belarus | 47 | 44 | 91
  India | 26 | 31 | 57

OUTCOME MEASURES:

1. Primary Outcome: To Achieve Clinical Remission in Subjects With Active Ulcerative Colitis (UC).
Description: Clinical remission defined as stool frequency score of 0, rectal bleeding score of 0, no urgency
Time Frame: 6 weeks
Population: ITT
Measure: Number; unit: participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
participants | 42 | 29
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority or Other; p = 0.069, Chi-squared

2. Secondary Outcome: Clinical Remission
Description: Clinical remission defined as a score of 0 for stool frequency, 0 for rectal bleeding and no urgency
Time Frame: 10 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
Participants | 57 | 30
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

3. Secondary Outcome: Endoscopic Remission
Description: Endoscopic remission is defined as a sigmoidoscopy score of 1 or less
Time Frame: 6 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
Participants | 64 | 35
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

4. Secondary Outcome: Endoscopic Remission
Description: Endoscopic remission is defined as a sigmoidoscopy score of 1 or less
Time Frame: 10 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
Participants | 73 | 52
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p = 0.010, Chi-squared

5. Secondary Outcome: Improvement
Description: Improvement is defined as a reduction of at least 3 points from baseline in the modified UC-DAI score. (minumum 3, maximum 7, higher absolute UC-DAI scores indicate more severe disease)
Time Frame: 6 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
Participants | 83 | 47
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Improvement
Description: as for outcome 5
Time Frame: 10 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 140 | 141
Participants | 88 | 57
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p < 0.001, Chi-squared

7. Post Hoc Outcome: To Achieve Clinical Remission in the Patient Population Confirmed by the Central Reader
Description: Clinical Remission, defined as stool frequency score of 0, rectal bleeding score of 0 and absence of urgency in subjects with adequate disease extent at baseline confirmed by central reading.
Time Frame: 6 weeks
Population: modified ITT, eligibility confirmed by central reader
Measure: Count of Participants; unit: Participants
Arm/Group | Mesalamin | Placebo
Number analyzed (Participants) | 107 | 87
Participants | 31 | 12
Statistical Analysis 1: Comparison: Mesalamin vs Placebo; Test type: Superiority; p = 0.011, Chi-squared

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | Mesalamin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/140 | 3/141
Other Adverse Events (participants affected / at risk) | 27/140 | 47/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamin (N=140) | Placebo (N=141)
Colitis ulcerosa (Gastrointestinal disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesalamin (N=140) | Placebo (N=141)
Monozytopenia (Investigations) | 5 (5) | 10 (10)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 7 (7)
Colitis ulcerosa (Gastrointestinal disorders) | 13 (13) | 30 (30)

LIMITATIONS AND CAVEATS:
Investigator endoscopy scores resultet in 31% patients with insuficient disease severity at baseline. Central reader scores were used for a post hoc analysis of the primary endpoint, including patients with pre-specified disease severity only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes